CLINICAL TRIAL: NCT06999083
Title: A Phase Ia, Randomized, Double-blind, Placebo-controlled, Single Dose-escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HB0043 in Healthy Adult Subjects
Brief Title: A Study to Evaluate Single-dose of HB0043 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: HB0043-HV-01-01
Record Dates: First submitted 2025-05-23; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: HB0043
MeSH Terms: interventions — Interleukin-1 Receptor Accessory Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- HB0043 dose group 1 (Active Comparator): HB0043 single dose
  Interventions: Drug: HB0043
- HB0043 dose group 2 (Active Comparator): HB0043 single dose
  Interventions: Drug: HB0043
- HB0043 dose group 3 (Active Comparator): HB0043 single dose
  Interventions: Drug: HB0043
- HB0043 dose group 4 (Active Comparator): HB0043 single dose
  Interventions: Drug: HB0043
- HB0043 dose group 5 (Active Comparator): HB0043 single dose
  Interventions: Drug: HB0043
- HB0043 dose group 6 (Active Comparator): HB0043 single dose
  Interventions: Drug: HB0043
- Matching placebo for each dose group (Placebo Comparator): placebo, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HB0043 — HB0043 Drug Product
  Other Names: recombinant humanized IgG1 bispecific antibody targeting both IL-17A and IL-36R.
  Arms: HB0043 dose group 1; HB0043 dose group 2; HB0043 dose group 3; HB0043 dose group 4; HB0043 dose group 5; HB0043 dose group 6
Drug: Placebo — Placebo
  Arms: Matching placebo for each dose group

SUMMARY:
The aim of this study is to investigate the safety and tolerability of HB0043 in healthy subjects following single-dose.

DETAILED DESCRIPTION:
This is a single-dose escalation study of HB0043 to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of HB0043.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following criteria to be eligible for study entry:

  1. Healthy male or female subjects age ≥ 18 and ≤ 55 years.
  2. Men and women of reproductive potential, willing to practice a highly effective method of birth control for the duration of the study and continuing for 6 months after receiving the last dose of drug administration. Highly effective methods of birth control include sexual abstinence (men, women); vasectomy or a condom (men) in combination with other barrier methods, hormonal birth control or IUD (women).
  3. Body Mass Index (BMI) ≥ 18 and ≤ 32 kg/m².
  4. No clinically significant findings in the medical history and physical examination.
  5. No clinically significant laboratory values (including urinalysis), unless the investigator considers any abnormality to not be clinically significant.
  6. Normal ECG, blood pressure, respiratory rate, temperature and heart rate, unless the investigator considers any abnormality to be not clinically significant.
  7. Informed consent must be obtained for all subjects enrolled into the study.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from study entry:

1. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disease.
2. Current or history of malignancy.
3. Family history of premature Coronary Heart Disease (CHD).
4. Treatment in the previous 3 months with any drug known to have a well-defined potential for toxicity to a major organ. Exposure to any prescription medication 14 days prior to randomization, to herbal remedies or over-the countermedications (except for the occasional use of acetaminophen [up to 2,000 mg per day]) 7 days prior to randomization.
5. Participation in another research with any investigational product within 28 days or 5 half-lives of the drug, whichever is greater, before screening.
6. Known allergy to biologics.
7. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing
8. Had a vaccination with a live attenuated vaccine within 1 months prior to dosing.
9. Subjects at risk for tuberculosis (TB), specifically subjects with:

   * Current clinical, radiographic or laboratorial evidence of active TB;
   * Positive interferon-γ release assay (IGRA) test.
10. Positive test at screening for any of the following infectious disease tests: Hepatitis B, surface antigen (HBsAg), Hepatitis C virus antibody (HCV Ab), Human immunodeficiency virus antibody (HIV Ab).
11. History of clinically significant opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia).
12. A helminth parasitic infection diagnosed within 6 months prior to screening that has not been treated with, or has failed to respond to, standard of care therapy.
13. Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to screening.
14. Presence of fever (body temperature >37.5°C) (e.g., a fever associated with a symptomatic viral or bacterial infection) within 2 weeks prior to the first dosing.
15. History of drug abuse within 1 year prior to screening, or use of soft drugs (such as marijuana) within 3 months prior to the screening, or hard drugs (such as cocaine, phencyclidine, and crack) within 1 year prior to screening. Positive drug screen (cocaine, methamphetamine, phencyclidine, and Tetrahydrocannabinol) at screening or Day -1.
16. History of regular alcohol consumption exceeding 14 drinks/week for female subjects or 21 drinks/week for male subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening. Positive Breath Alcohol Test at screening or Day -1.
17. Current cigarette smoker (cigarettes or e-cigarettes) who smoke over 5 cigarettes/day within 3 months prior to screening.
18. Mental condition rendering the subject incapable of understanding the nature, scope, and possible consequences of the study.
19. Pregnant or Breasting feeding subject. Women with positive pregnancy test (hCG). Or subjects who plan to donate sperms or eggs, from dosing until at least 6 months after last dose of investigational medicine.
20. Adults under guardianship and people with restriction of freedom by administrative and legal decisions.
21. Unlikely to comply with the clinical study protocol, e.g. uncooperative attitude, inability to return for followed-up visit, and improbability of completing the study.
22. Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative there of directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-06-03 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with drug related adverse events (AEs) | Up to 1200 hours
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational drug

SECONDARY OUTCOMES:
Cmax | Up to 1200 hours
  The maximum measured concentration of the analysis in plasma.
AUC0-infinity | Up to 1200 hours
  The area under the concentration-time curve of the analysis in plasma over the time interval from 0 extrapolated to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Millie Wang, Principal Investigator — New Zealand Clinical Research
Locations (1):
- New Zealand Clinical Research , Grafton, Auckland, 3 Ferncroft Street,, Auckland, Grafton, New Zealand

IPD SHARING:
Plan to Share IPD: No